CLINICAL TRIAL: NCT05981209
Title: Phase 1b Study to Assess Safety and Efficacy of Elotuzumab, CC-92480, and Dexamethasone in Relapsed/Refractory Myeloma After CD38- and BCMA-Targeted Therapies
Brief Title: Elotuzumab, CC-92480, and Dexamethasone for the Treatment of Relapsed or Refractory Myeloma After CD38- and BCMA-Targeted Therapies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abdullah Khan (Other)
Responsible Party: Sponsor-Investigator, Abdullah Khan, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22207; NCI-2023-05518 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; elotuzumab; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (elotuzumab, CC-92480, dexamethasone) (Experimental): Patients receive elotuzumab IV on days 1, 8, 15, and 22 of cycles 1 and 2 and then on day 1 of each subsequent cycle. Patients also receive CC-92480 PO on days 1-21 of each cycle and dexamethasone IV or PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo an ECHO during screening and undergo MRI, CT, or x-ray imaging during screening and on study as clinically indicated. Patients also undergo blood sample collection as well as bone marrow biopsy and aspiration during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Echocardiography; Biological: Elotuzumab; Procedure: Magnetic Resonance Imaging; Biological: Mezigdomide; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; Empliciti; HuLuc-63; HuLuc63; PDL-063; PDL063
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Mezigdomide — Given PO
  Other Names: BMS 986348; BMS-986348; BMS986348; CC 92480; CC-92480; CELMoD CC-92480; Cereblon E3 Ligase Modulation Drug CC-92480; Cereblon E3 Ubiquitin Ligase Modulating Agent CC-92480; Cereblon Modulator CC-92480
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of CC-92480 in combination with elotuzumab and dexamethasone in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that does not respond to treatment or has not responded to previous treatment (refractory). Multiple myeloma (MM) remains the second most common hematologic malignancy in the United States. A number of therapies have been approved for patients with MM, including CD38- and B-cell maturating antigen (BCMA)-targeted therapies (antibody and plasma cell treatments that help the body's immune system to kill cancer cells); however, patients will often relapse and become refractory to these therapies. Because of this, it is important to identify effective treatment options for patients progressing on anti-CD38 therapy and BCMA-directed therapies. Elotuzumab is a humanized IgG1 monoclonal antibody, which is a type of protein that can bind to other target cells to prevent them from working the way they should or cause them to act differently. Elotuzumab works by targeting a protein called SLAMF7, which is present on myeloma cells, and makes it easier for the immune system to target the cancer. CC-92480 works by binding to a protein called CRBN that triggers the breakdown of proteins: Ikaros and Aiolos, leading to cell death in multiple myeloma cells. Dexamethasone is a synthetic adrenocortical steroid, or steroid normally naturally made by the adrenal gland in the brain which has been produced in a laboratory, that helps to regulate the amount of different chemicals and water that are being processed by the kidneys. It is also used in patients with myeloma to help treat their disease. The combination of CC-92480 with elotuzumab and dexamethasone may be a safe and effective treatment when given to patients with relapsed or recurrent MM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of elotuzumab, mezigdomide (CC-92480), and dexamethasone (E480d) in patients with relapsed/refractory multiple myeloma (RRMM) who have received >= 2 prior regimens including CD38- and BCMA-targeted therapies.

SECONDARY OBJECTIVES:

I. Determine the time to response (TTR), the duration of response (DOR), very good partial response [VGPR] or better and complete response [CR] rates, progression free survival (PFS) at 1 year, and overall survival (OS) at 1 year.

II. Check minimal residual disease (MRD) negativity rates by next generation sequencing in patients who are suspected of attaining a complete response (CR).

III. Correlative studies will include changes in lymphocyte subsets with therapy, immunophenotype of MM cells, and expression of CRBN, Ikaros, and Aiolos.

IV. Quality of life (QOL) will be assessed.

OUTLINE: This is a dose-escalation study of CC-92480, followed by a dose-expansion study.

Patients receive elotuzumab intravenously (IV) on days 1, 8, 15, and 22 of cycles 1 and 2 and then on day 1 of each subsequent cycle. Patients also receive CC-92480 orally (PO) on days 1-21 of each cycle and dexamethasone IV or PO on days 1, 8, 15, and 22 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may undergo an echocardiography (ECHO) during screening and undergo magnetic resonance imaging (MRI), computed tomography (CT), or x-ray imaging during screening and on study as clinically indicated. Patients also undergo blood sample collection as well as bone marrow biopsy and aspiration during screening and on study.

After completion of study treatment, patients are followed up at 30 and 60 days and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with evidence of relapsed or refractory disease as defined by International Myeloma Working Group (IMWG) criteria and measurable disease as defined by any of the following:

  * Serum M-protein >= 1.0 g/dl
  * Urine monoclonal protein >= 200 mg/24h
  * Involved free light chain (FLC) level >= 10mg/dl (>= 100mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
* Patients must have had at least 2 prior lines of therapy including lenalidomide, proteasome inhibitor (PI), anti-CD38 directed antibody, and BCMA-targeted therapy

  * Prior elotuzumab is permitted but patients with progressive disease (PD) as best reponse on elotuzumab are excluded; at least 6 months must have lapsed from prior elotuzumab exposure
* Patients must have hemoglobin >= 7g/dL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 70,000/uL

  * If plasma cell percentage on bone marrow biopsy aspirate or core is > 30%, platelet requirement will be adjusted to 50,000/ul
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/alkaline phosphatase < 2.5 x the ULN
* Calculated creatinine clearance of >= 45ml/min using Modification of Diet in Renal Disease (MDRD) formula
* Left ventricular ejection fraction >= 30%; baseline echocardiography (ECHO) is not required if ECHO was done within the preceding one year and patients do not have new signs/symptoms suggestive of heart failure
* No uncontrolled arrhythmias
* No New York Heart Association class III-IV heart failure
* 12-lead electrocardiogram (ECG) with QT interval calculated by Fridericia formula (QTcF) interval of =< 470 msec
* Patient must be able to swallow capsule or tablet
* Patients must provide informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of < 2
* Women of child bearing potential (WOCBP) must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing and continue to 6 months after study treatment ending. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy
* Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy
* A negative pregnancy test will be required for all WOCBP within 24 hours before starting treatment drugs
* Breast feeding is not permitted while taking study drug, during dose interruptions, and for 28 days after the last dose of study drug.
* Females should refrain from ova donation during this time and continue for 28 days after study treatment ending.
* Male patients must agree to use an adequate method of contraception (latex or synthetic condom) while taking the study drug, during dose interruptions, and up to 28 days following the last dose of study drug
* Criteria also applies to azoospermic males and those who have had vasectomy
* Males should refrain from sperm donation during this time and continue for 6 months after study treatment ending

Exclusion Criteria:

* Patients with Waldenstrom macroglobulinemia, primary amyloid light chain (AL) amyloidosis, primary plasma cell leukemia, or polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma cell disorder, skin changes (POEMS) syndrome

  * Patients with secondary plasma cell leukemia are permitted
* Patients with peripheral neuropathy > National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 2, or grade 2 peripheral neuropathy with pain
* Patients receiving concurrent corticosteroids at the time protocol therapy is initiated other than for physiologic maintenance treatment
* Concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of the study drugs
* Patients with history of anaphylaxis or hypersensitivity to elotuzumab, lenalidomide, or pomalidomide
* Concurrent use of strong CYP3A modulators ≤ 2weeks; concurrent use of proton-pump inhibitors =< 1 weeks prior to started CC-92480; potassium competitive acid blockers ≤ 2days prior to starting CC-92480
* Unacceptable respiratory risk factors defined by any one of the following criteria:

  * Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) less than 50% of predicted normal
  * Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Unacceptable cardiac risk factors defined by any of the following criteria:

  * Left ventricular ejection fraction < 30%
  * Complete left bundle branch, bifascicular block or clinically significant abnormal electrocardiogram (EKG) finding at screening
  * A prolongation of QT interval on screening ECG as defined by repeated demonstration of a QTc interval > 470 msec using Fridericia's QT correction formula; a family history of long QT syndrome
  * Myocardial infarction within 6 months
  * Unstable angina
* Patients who have received targeted or investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is shorter) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with active hepatitis B (defined as hepatitis B surface antigen [HBsAg]+); hepatitis b virus (HBV) screening is required prior to beginning therapy

  * Patients with prior hepatitis B vaccine are permitted (defined as HBsAg-, hepatitis B virus surface antibody [anti-HBs]+, hepatitis B virus core antibody [anti-HBc]-)
  * Non-active hepatitis B (HBsAg-, anti-HBs+, anti-HBc+) may only be enrolled following approval by the sponsor after consideration of risk of reactivation (additional screening and monitoring for hepatitis B and consultation with a liver disease specialist may be required)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention, other than non-melanoma skin cancer and carcinoma in situ of the cervix or breast, should not be enrolled
* Patients with a history of gastrointestinal surgery or other procedure that might, in the opinion of the investigator(s), interfere with the absorption or swallowing of the study drugs
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The recommended phase 2 dose of mezigdomide (CC-92480) in combination with elotuzumab and dexamethasone | Up to 28 days (Cycle 1)
  The dose limiting toxicity (DLT) will be defined as one or more of the following toxicities considered to be at least possibly related to the study drug, occurring during cycle 1 of therapy. Furthermore, inability to take >= 75% of the planned CC-92480 doses, or receive cycle 2 day 1 doses due to a drug-related adverse event occurring in cycle 1 will be considered a DLT.
Incidence of adverse events | Up to 2 years
  Adverse events and toxicities of the combination regimen will be summarized using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicities will be assessed overall, as well as by dose level. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. The incidence of severe (grade 3+) adverse events or toxicities will be described. Will also assess tolerability of the regimen through assessing the number of patients who required dose modifications and/or dose delays. In addition, will capture the proportion of patients who go off treatment due to adverse reactions. All patients who have received at least one dose of any of the study regimen will be evaluable for toxicity.

SECONDARY OUTCOMES:
Time to progression (TTP) | From start of treatment until objective tumor progression; with death as a competing risk, assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. For TTP, cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks.
Time to response (TTR) | From start of treatment until measurement criteria are first met for PR, very good partial response (VGPR), or complete response (CR) (whichever status is recorded first), assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. For TTR, cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks
Duration of response (DOR) | From the time measurement criteria are first met for partial response or better (whichever status is recorded first) until the first date of progressive disease or death, assessed at 1 year
  DOR will be computed for subjects whose best response is either PR, VGPR, or CR. Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. DOR will be analyzed using the Kaplan-Meier method. The probability of survival and median DOR will be calculated together with 95% CIs, and log-rank test will be used for the comparison between patient subgroups.
Very good partial response (VGPR) or better rates | From start of treatment until disease progression or death, assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. VGPR will be analyzed using the Kaplan-Meier method. The probability of survival and median DOR will be calculated together with 95% CIs, and log-rank test will be used for the comparison between patient subgroups.
Complete Response (CR) | From start of treatment until disease progression or death, assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. CR will be analyzed using the Kaplan-Meier method. The probability of survival and median DOR will be calculated together with 95% CIs, and log-rank test will be used for the comparison between patient subgroups.
Progression free survival (PFS) | From start of treatment until disease progression or death, assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. PFS will be analyzed using the Kaplan-Meier method. The probability of survival and median PFS will be calculated together with 95% CIs, and log-rank test will be used for the comparison between patient subgroups.
Overall survival (OS) | From start of treatment to the date of his or her death, assessed at 1 year
  Primary evaluation of antitumor activity of study treatment will be assessed according to IMWG response criteria. OS will be analyzed using the Kaplan-Meier method. The probability of survival and median OS will be calculated together with 95% CIs, and log-rank test will be used for the comparison between patient subgroups.
Minimal residual disease (MRD) | At final study visit, up to 2 years
  Planned for patients suspected of attaining CR. MRD negativity is associated with superior outcomes compared to MRD positivity.
Changes in lymphocyte subsets with therapy | Up to 2 years
  Changes in expression of these markers across time will be explored by dose level graphically. Relationships between changes in lymphocyte subsets, total number and ratio of regulatory T cells will be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries, compared using Mann-Whitney test or Fisher exact test depending on the data type of expression data.
Changes in immunophenotype of multiple myeloma cells | Up to 2 years
  Correlative studies including the changes in expression of these markers across time will be explored by dose level graphically.
Changes in expression of CRBN, Ikaros, and Aiolos with therapy | Up to 2 years
  Changes in expression of these markers across time will be explored by dose level graphically.
Quality of life (QOL) | At baseline and monthly until study completion, up to 2 years
  Measured with the Patient-Reported Outcomes Measurement Information System Global 10 Quality of Life Survey and The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma20. A repeated measures linear mixed model will be fit to all QOL scores. The model will include all time points (baseline as reference session 0 and 1-6 or higher for each monthly measure), and a patient-level random effect. A p-value for the difference between baseline QOL and QOL at the end of the study will be obtained from the model, and if the positive difference with p-value is < 0.05 QOL will be seen as improved.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Khan, MBBS, MSc, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu